CLINICAL TRIAL: NCT02688660
Title: MRI Markers of Outcome After Severe Pediatric Traumatic Brain Injury (TBI)
Brief Title: MRI Markers of Outcome After Severe Pediatric TBI
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0185; R01NS092870 (NIH); A536700 (Other: UW Madison); PEDIATRICS-GEN (Other: UW Madison); Protocol Version 8/28/2019 (Other: UW Madison)
Record Dates: First submitted 2016-01-29; First posted 2016-02-23 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-04

CONDITIONS: Brain Injuries
Keywords: Pediatrics; Neuroimaging
MeSH Terms: conditions — Brain Injuries | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ADAPT Study Population: This cohort will be subjects from the ADAPT study who had an acute MRI scan which has been uploaded into the ADAPT database from all participating sites.
- Follow-Up MRI: This cohort will include patients from ADAPT sites who choose to participate in this option and obtain a follow-up MRI approximately 1 year after the TBI.
  Interventions: Other: MRI Scans
- Healthy Controls: This cohort will have one MRI to be used in comparison of the above cohorts.
  Interventions: Other: MRI Scans

INTERVENTIONS:
Other: MRI Scans
  Groups: Follow-Up MRI; Healthy Controls

SUMMARY:
Traumatic brain injury (TBI) is the leading cause of death or disability in children. Each year in the United States, pediatric TBI results in an estimated 630,000 emergency room visits, 58,900 hospitalizations, and 7000 deaths. The incidence of long-term disability after severe TBI is high, with over 60% of children requiring educational or community based supportive services 12 months post-injury. Over 5,000 children require inpatient rehabilitation after TBI each year and an estimated 145,000 US children are currently living with disabilities after a severe TBI. Hospital costs for the acute treatment of children with TBI are estimated at ~$2.6 billion each year, while the gross annual costs accounting for long-term care and lost productivity approach $60 billion. Therefore, pediatric TBI is a major public health concern and new ways to diagnose and treat TBI are urgently needed.

DETAILED DESCRIPTION:
Severe pediatric TBI results in a range of neurocognitive and behavioral deficits with resultant impact on school performance, social functioning, and quality of life. Sixty percent of children suffer from long-term functional impairments after severe TBI, and more than 40% demonstrate deficits in multiple cognitive and psychological domains. Importantly, a recent meta-analysis revealed that rather than catching up to their peers in these domains, children with severe TBI fall further behind over time. These deficits in cognitive and emotional function have a major impact on the child's quality of life after a TBI. A large study recently reported that severe TBI patients demonstrated lower quality of life than children undergoing active treatment for cancer. Considerable variation exists in the severity of impairment within each cognitive domain from patient to patient, likely relating to the mechanism of injury, the type and location of lesion, patient age, and pre-morbid functioning among other factors. While clinical scales such as the Glasgow Coma Scale (GCS) are useful for assessing injury severity and may provide general prognostic information, they are insufficient to identify risk for specific cognitive deficits. Identifying predictors of impairment within specific domains would aid in directing rehabilitation strategies towards at-risk cognitive domains, thereby improving long-term function and quality of life.

The investigators are partnering with an ongoing pediatric TBI trial (ADAPT Trial: Approaches and Decisions in Acute Pediatric TBI) and will also be enrolling past UW patients and healthy controls. Consistency in timing of follow-up scans, large sample size and access to the ADAPT Trial injury severity data and neuropsychological testing will give this study unprecedented power to assess the relationship between early MRI findings and subsequent atrophy, white matter injury, network connectivity changes and neurocognitive and behavioral impairments.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 Subjects:

* Children 0 through < 18 years of age
* Diagnosis of severe TBI (defined as a Glasgow Coma Scale (GCS) score less than or equal to 8)
* Had an intracranial pressure (ICP) monitor as part of standard care

Aims 2 & 3 Subjects:

* Children 9 through < 18 years of age with severe TBI
* Consent for a follow-up MRI within 10 years of the time of TBI

Controls:

* Healthy children greater than or equal to 9 and < 18 years of age.

Exclusion Criteria:

* TBI & controls:
* Anyone unable to tolerate a non-sedated MRI

Controls:

* Any history of head injury resulting in loss of consciousness
* Standard contraindications to MRI (metallic implants, implanted electronic devices, pregnancy, etc.).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients who have experienced TBI and had an acute MRI scan and those who participate in the prospective phase and obtain a follow-up MRI. Healthy controls will also be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Cerebral Atrophy | 1 year
  Global and regional cerebral atrophy will be assessed using MRI
White matter fractional anisotropy | 1 year
  Fractional Anisotropy will be assessed using Diffusion Tensor MRI
Brain network connectivity | 1 year
  Network connectivity will be assessed using resting-state functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ferrazzano, MD, Principal Investigator — University of Wisconsin, Madison
Locations (21):
- United States (18):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - UC San Diego Health Sciences Center, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - American Family Children's Hospital (AFCH), Madison, Wisconsin
- The Royal Children's Hospital, Melbourne, Victoria, Australia
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham, England
  - University Hospital Southampton, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bigler ED, Abildskov TJ, Petrie J, Farrer TJ, Dennis M, Simic N, Taylor HG, Rubin KH, Vannatta K, Gerhardt CA, Stancin T, Owen Yeates K. Heterogeneity of brain lesions in pediatric traumatic brain injury. Neuropsychology. 2013 Jul;27(4):438-51. doi: 10.1037/a0032837. PMID 23876117
- [Background] Tasker RC, Westland AG, White DK, Williams GB. Corpus callosum and inferior forebrain white matter microstructure are related to functional outcome from raised intracranial pressure in child traumatic brain injury. Dev Neurosci. 2010;32(5-6):374-84. doi: 10.1159/000316806. Epub 2010 Sep 8. PMID 20829579
- [Background] Birn RM, Shackman AJ, Oler JA, Williams LE, McFarlin DR, Rogers GM, Shelton SE, Alexander AL, Pine DS, Slattery MJ, Davidson RJ, Fox AS, Kalin NH. Evolutionarily conserved prefrontal-amygdalar dysfunction in early-life anxiety. Mol Psychiatry. 2014 Aug;19(8):915-22. doi: 10.1038/mp.2014.46. Epub 2014 May 27. PMID 24863147
- [Background] Yue JK, Vassar MJ, Lingsma HF, Cooper SR, Okonkwo DO, Valadka AB, Gordon WA, Maas AI, Mukherjee P, Yuh EL, Puccio AM, Schnyer DM, Manley GT; TRACK-TBI Investigators. Transforming research and clinical knowledge in traumatic brain injury pilot: multicenter implementation of the common data elements for traumatic brain injury. J Neurotrauma. 2013 Nov 15;30(22):1831-44. doi: 10.1089/neu.2013.2970. Epub 2013 Sep 24. PMID 23815563
- [Background] Beers SR, Wisniewski SR, Garcia-Filion P, Tian Y, Hahner T, Berger RP, Bell MJ, Adelson PD. Validity of a pediatric version of the Glasgow Outcome Scale-Extended. J Neurotrauma. 2012 Apr 10;29(6):1126-39. doi: 10.1089/neu.2011.2272. Epub 2012 Apr 10. PMID 22220819
- [Background] McCauley SR, Wilde EA, Anderson VA, Bedell G, Beers SR, Campbell TF, Chapman SB, Ewing-Cobbs L, Gerring JP, Gioia GA, Levin HS, Michaud LJ, Prasad MR, Swaine BR, Turkstra LS, Wade SL, Yeates KO; Pediatric TBI Outcomes Workgroup. Recommendations for the use of common outcome measures in pediatric traumatic brain injury research. J Neurotrauma. 2012 Mar 1;29(4):678-705. doi: 10.1089/neu.2011.1838. Epub 2011 Aug 24. PMID 21644810
- [Background] Alexander AL, Lee JE, Lazar M, Field AS. Diffusion tensor imaging of the brain. Neurotherapeutics. 2007 Jul;4(3):316-29. doi: 10.1016/j.nurt.2007.05.011. PMID 17599699